CLINICAL TRIAL: NCT03416322
Title: Impact of Water-assisted Colonoscopy vs Second Forward View Examination of the Right Colon on Adenoma Detection
Brief Title: Water-assisted Colonoscopy vs Second Forward View Examination of the Right Colon on Adenoma Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Denise Peixoto Guimarães, MD, PhD, Barretos Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BarretosCH-20173
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Adenoma; Colorectal Cancer
Keywords: Adenoma; Adenoma detection rate; Colorectal cancer
MeSH Terms: conditions — Adenoma; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Clinical, prospective and comparative, randomized study. Patients referred to the Endoscopy Department of the Barretos Cancer Hospital from August 2017 to August 2018 will be invited to participate in the study, with an indication of performing a diagnostic colonoscopy for high-risk CCR screening (Lynch and Li Fraumeni Syndrome) or who are in post-polypectomy follow-up.
  After agreeing and signing the Informed Consent Term (ICF), the included patients will be divided into two groups. The first group will be submitted to the technique of "second right frontal view of the right colon" (SEVF), which consists in reexamining the right colon after reaching the hepatic angle on colonoscope withdrawal. The second group will be submitted to the "Underwater" technique, which consists in evaluating the right colon after this segment has been cleaned with water, injected water and aspirated after. During aspiration of water, the colon will be examined.
Who Masked: Participant
Masking Description: Randomization of participants will be done in a 1:1 ratio, with the random sequence in blocks 2, 4 and 6. The sequence of treatments within the blocks and the block sequence will be randomized. For this randomization, the REDCap platform will be used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Second Examination of the right colon (No Intervention): Second forward view examination of the right colon once the right colon (cecum to hepatic flexure) has been examined
- Water exchange (Experimental): Water infusion during colonoscope insertion in the right colon (from hepatic flexure to cecum) and remove water during withdrawn ("Exchange method").
  Interventions: Other: Water exchange

INTERVENTIONS:
Other: Water exchange — Infusion and remove water during inertion and withdrawal of colonoscope
  Arms: Water exchange

SUMMARY:
Introduction and objectives: The adenoma detection rate (ADR) has been investigated as a formal method in the evaluation of a trainee or resident physician. Several studies have suggested that water-assisted colonoscopy methods increase the ADR, especially in the right colon, when compared to air-insufflated methods alone. The objective of this study is to compare the adenoma detection rates between the techniques of the second frontal view examination and "Underwater" examination by residents, supervised by a senior endoscopist.

Patients and methods: This is a prospective, comparative and randomized clinical trial. The patients referred to the Cancer Hospital of Barretos for colonoscopy, and who agreed with the study, were divided into two groups, one with the use of water and the other only with air insufflation. The primary endpoint of this study is to compare adenoma detection rate. Secondary outcomes were withdrawal time, proportion of intubation of the cecum, preparation of the colon, and number of previously performed colonoscopies in the ADR in both techniques.

DETAILED DESCRIPTION:
Introduction Colorectal cancer (CRC) is one of the most common cancers in the world. In Brazil, it is the second most incident tumor in women and the third in men. Colonoscopy is considered the gold standard test for colorectal cancer screening through the detection and removal of adenomas or detection of early cancers. However, this protection is not perfect and even less effective in the right colon (cecum and ascending colon) when compared to the distal colon, which leads to underdiagnosis of neoplasias and precursor lesions (eg adenomas). In this context, the performance and quality of colonoscopy play an important role in minimizing colonoscopy deficiencies. The American Society for Gastrointestinal Endoscopy (ASGE) determines three indispensable indicators for measuring the quality of colonoscopy: cecal intubation (≥95% in screening colonoscopies), adenoma detection rate (ADR) (≥25% in men and women, on screening colonoscopies) and withdrawal time (≥6 minutes on screening, negative colonoscopies).

In addition, for a better detection of lesions, it is necessary that the assessed colonic segment be cleaned of residues, and, therefore, proper colonic preparation is one of the quality items of the examination. Inadequate preparation impairs the detection of polyps and flat lesions, increases the time of the examination, increases the chances of complications and the costs of colonoscopy. One way to measure the quality of bowel preparation is the Boston Intestinal Prepare Scale. This scale uses a classification from 0 to 9 evaluating the preparation in three segments (right colon, transverse colon and left colon) after cleaning maneuvers. The score ranges from 0 (poor preparation) to 9 (excellent preparation).

In order to increase the quality of the colonoscopic examinations by increasing the ADR and reducing the incidence of the interval CRC, some methods have been investigated, including the Second Foward View Examination of the right-side colon (SFVE) and examination with Water Aid or Underwater colonoscopy (UW).

The first method is to evaluate the right colon with air and, upon reaching the hepatic flexsure, return to the cecum and re-evaluate the colonic segment. The second method, is to evaluate the right colon by inserting the colonoscope with the device completely immersed in water and withdrawn from the colonoscope with air after complete aspiration of the water, also known as the "Exchange method". The principle is that water cleans the colon and allows an increase of the image that is visualized by the colonoscope, and in that way, would improve the visualization of the mucosa.

Clark et al. demonstrated that, after performing SFVE, additional adenomas were found in 43 of 280 patients evaluated (15.4%, p <0.05) and the overall adenoma detection rate increased by 3.2% (p <0.05). The ADR in the right colon increased by 6.7% (p <0.05).

A retrospective study conducted by Leung et al. demonstrated that the UW technique increased the ADR in the right colon - at least one adenoma of any size was detected in 26.8% of patients in the air-evaluated group and in 34, 9% of patients in the group evaluated with water.

The two techniques showed to increase the ADR. Both are easy to carry out, do not require extra training or additional equipment, and have low cost. However, the impact of water exchange method colonoscopy on adenoma detection rate have not benn completely calrified. Further there is no evidence in the literature comparing these two techniques.

During colonoscopy learning curve, objective criteria are increasingly being suggested to assess the competence of "trainees". Traditionally, this evaluation is made by the number of procedures performed by them, but recently other criteria such as quality indicators, the ADR and intubation of the cecum have been investigated as formal methods in the evaluation of a trainee or resident. During the endoscopy residency in Barretos Cancer Hospital, surveillance colonoscopies are performed by residents supervised by the senior endoscopistThere is currently no evaluation of the colonoscopy technique performed by the resident. In addition, there is no evaluation of the ADR during the learning curve of the endoscopy resident in our department.

Justification The need to ensure adequate ADR among endoscopy residents. Absence of studies comparing UW and SEVF techniques of the right colon for the adenoma detection rate.

Primary objective To compare the ADR between combined SEFV and UW techniques in the right colon in patients undergoing colonoscopy for high-risk screening, diagnosis and follow-up after polypectomy, performed by residents supervised by a senior endoscopist.

Secondary objectives To estimate the association between withdrawal time, proportion of independent intubation of the cecum, preparation of the colon and the number of previously performed colonoscopies in the ADR in both techniques previously performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing diagnostic colonoscopy and surveillance colonoscopy

Exclusion Criteria:

* Contraindication for performing the endoscopic procedure.
* Refusal to provide inform consent.
* Past history of partial colectomy, familial adenomatous polyposis, inflammatory bowel disease, coagulopathy or thrombocytopenia.
* Incomplete colonoscopy
* Inadequate bowel preparation
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | up to 12 months
  Proportion of individuals with at least one adenoma

SECONDARY OUTCOMES:
Detection rate of any clinically significant lesion | up to 12 months
  Proportion of participants with at least one clinically significant lesion (adenoma, serrated or cancer)
Detection rate of serrated adenoma | up to 12 monthas
  Proportion of participants with at least one serrated adenoma total and per resident
Colonoscopy completion rate per resident | up to 12 months
  Proportion of complete colonoscopies per resident, independently of the senior examiner
Cecal intubation time | up to 12 months
  Time it takes from anal insertion ti the time the tip of colonoscope in the the cecum
Colonoscopy withdrawal time | up to 12 months
  time it takes to withdraw colonoscope
Boston Intestinal Preparation Scale | up to 12 months
  Proportion of participants with boston scale grade

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Guimaraes, Barretos, São Paulo, Brazil